CLINICAL TRIAL: NCT01945762
Title: European, Observational, Prospective Study to Evaluate the Benefit/Risk of Vandetanib in RET Mutation Negative and Positive Patients With Symptomatic, Aggressive, Sporadic, Unresectable, Locally Advanced/Metastatic Medullary Thyroid Cancer
Brief Title: Observational Study to Evaluate Vandetanib in RET -/+ Patients With Metastatic Medullary Thyroid Cancer
Acronym: Caprelsa104
Status: Completed | Type: Observational
Sponsor: Genzyme, a Sanofi Company (Industry)
Collaborators: Worldwide Clinical Trials (Other)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Other Study IDs: D4200C00104; OBS14778 (Other: Sanofi)
Record Dates: First submitted 2013-09-10; First posted 2013-09-19 (Estimated); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Symptomatic, Aggressive, Sporadic, Unresectable, Locally; Advanced/Metastatic Medullary Thyroid Cancer (MTC)
Keywords: RET Mutation; DIagnostics; Medullary Thyroid Cancer; MTC
MeSH Terms: conditions — Aggression; Carcinoma, Medullary | interventions — vandetanib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1. patient cohorts (40 patients/cohort): RET positive patient cohorts
  Interventions: Drug: Vandetanib 300 mg
- 2. patient cohorts (40 patients/cohort): RET negative patient cohorts
  Interventions: Drug: Vandetanib 300 mg

INTERVENTIONS:
Drug: Vandetanib 300 mg — Vandetanib commercial tablets
  Other Names: ZD6474, CAPRELSA

SUMMARY:
This is a European multinational, multicenter, non-interventional (observational) and prospective study. It is carried on to confirm in real life conditions the benefit/risk of vandetanib (CAPRELSA™) 300 mg, both in RET negative and RET positive patients with symptomatic, aggressive, sporadic, unresectable, locally advanced/metastatic MTC.

DETAILED DESCRIPTION:
This is a multinational, multicenter, non-interventional (observational) and prospective study. European countries where vandetanib is on the market will participate in the study.

This study is being conducted to fulfil the specific obligation post-authorisation measure for the conditional marketing authorisation. It is carried on to confirm in real life conditions the benefit/risk of vandetanib (CAPRELSA™) 300 mg, both in RET negative and RET positive patients with symptomatic, aggressive, sporadic, unresectable, locally advanced/metastatic MTC. The clinical benefit of vandetanib (CAPRELSA™) 300 mg has previously been established in a clinical trial (Study 58) on the basis of a clinically and statistically significant advantage in progression free survival (PFS) which was supported by a high response rate and substantial duration of response.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent 2. Male or female aged 18 years or above 3. Histological diagnosis of MTC 4. Patients with symptomatic and aggressive sporadic MTC, who have unresectable, locally advanced/metastatic disease. (The factors considered by the investigator to determine a patient's disease to be symptomatic and aggressive will be recorded in the CRF). 5. Measurable disease:

* assessment confirmed within the 12 weeks previous to start of treatment, and
* defined according to RECIST 1.1: at least one lesion, not irradiated, that can be accurately measured as ≥10 mm in the longest diameter (except lymph nodes which must have short axis ≥15 mm) with CT or MRI and which is suitable for accurate repeated measurements. Measurable lesions with calcifications should not be assessed as target lesions unless no other measurable lesion is available. 6. Known definite RET mutation status (definition according to section 3.2). The status should be:
* for patients prescribed with vandetanib: positive or negative
* for patients not prescribed with vandetanib: negative RET mutation status must be determined from a tumour sample obtained within 18 months prior to enrollment. It is strongly recommended that a tissue sample obtained within 6 months prior to enrolment is used. 7. For patients newly prescribed vandetanib 300 mg, the prescription should be issued according to marketing authorisation and following the vandetanib Summary of Product Characteristics (SmPC) (Appendix B). The starting dose could be reduced to 200 mg in patients with moderate renal impairment

  * Exclusion criteria

    1. Current or planned inclusion/participation in a clinical trial
    2. Patients already receiving vandetanib or who have received vandetanib for their MTC before the study first visit
    3. Contraindications according to the vandetanib SmPC (not applicable for patients who do not receive vandetanib): (a) Patients with a QT interval corrected for heart rate (QTc) interval over 480 msec: (i) Congenital long QT syndrome (ii) Concomitant use of vandetanib with the following medicinal products known to also prolong the QT interval and / or induce Torsades de pointes: Arsenic, cisapride, erythromycin intravenous (IV), toremifene, mizolastine, moxifloxacin, Class I A and III antiarrhythmics (b) Currently pregnant or breast feeding (c) Hypersensitivity to the active substance or to any of the excipients (d) Severe renal impairment: creatinine clearance < 30 ml/minute calculated by Cockcroft-Gault formula. (See Appendix D). (e) Serum bilirubin greater than 1.5 x the upper limit of reference range (ULRR) (f) Potassium, magnesium or calcium outside the normal laboratory range

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Symptomatic, Aggressive, Sporadic, Unresectable, Locally Advanced/Metastatic Medullary Thyroid Cancer (MTC)
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2014-02-17 (Actual); Primary Completion 2020-06-18 (Actual); Study Completion 2020-06-18 (Actual)

PRIMARY OUTCOMES:
Assessment of Objective Response Rate | From enrollment until study completion, assessed up to 38 months
  Assessment of Objective Response Rate [using Response Evaluation Criteria In Solid Tumours (RECIST) 1.1]
Assessment of Disease control rate | From enrollment until study completion, assessed up to 38 months
  Assessment of Disease control rate [using Response Evaluation Criteria In Solid Tumours (RECIST) 1.1]
Assessment of Duration of Response | From enrollment until study completion, assessed up to 38 months
  Assessment of Duration of Response (using RECIST 1.1)
Assessment of Progression Free Survival | From enrollment until study completion, assessed up to 38 months
  Assessment of Progression Free Survival (using RECIST 1.1)
Evaluation of Safety by assessment of QTc prolongations | From enrollment until study completion, assessed up to 38 months
  Assessment of QTc prolongations
Evaluation of Safety by assessment of Adverse Events | From enrollment until study completion, assessed up to 38 months
  Assessment of Adverse Events
Evaluation of Safety by assessment of vital signs | From enrollment until study completion, assessed up to 38 months
  Assessment of Vital signs
Evaluation of Safety by assessment of laboratory data | From enrollment until study completion, assessed up to 38 months
  Assessment of Laboratory data

SECONDARY OUTCOMES:
Patient Characteristics | From enrollment until study completion, assessed up to 38 months
  Patient demographics and medical history / Disease characteristics / Death / Treatment information

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (8):
- investigational Site Belgium, Belgium, Belgium
- investigational Site France, France, France
- investigational Site Germany, Germany, Germany
- investigational Site Italy, Italy, Italy
- investigational Site Luxembourg, Luxembourg, Luxembourg
- investigational Site Netherlands, Netherlands, Netherlands
- investigational Site Spain, Spain, Spain
- investigational Site United Kingdom, United Kingdom, United Kingdom

REFERENCES:
- See also: OBS14778 clinical study synopsis and addendum — http://catalogues.ema.europa.eu/node/3055/methodological-aspects#darwin-documents